CLINICAL TRIAL: NCT01986556
Title: A Phase 1, Randomized, Open-Label, Crossover Study in Healthy Adult Male Subjects to Assess the Relative Bioavailability of Lesinurad Tablets Manufactured at Two Different Sites
Brief Title: Lesinurad Tablet Relative Bioavailability
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ardea Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RDEA594-129
Record Dates: First submitted 2013-11-12; First posted 2013-11-18 (Estimated); Last update posted 2014-09-22 (Estimated); Status verified 2014-09

CONDITIONS: Healthy
MeSH Terms: interventions — lesinurad

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Lesinurad 400 mg Fasted (Site 1 and Site 2, Lot A) (Experimental): Day 1: Lesinurad 400 mg (Site 1 or Site 2, Lot A) Day 5: Lesinurad 400 mg (Site 1 or Site 2, Lot A)
  Interventions: Drug: Lesinurad 400 mg (Site 1); Drug: Lesinurad 400 mg (Site 2, Lot A)
- Lesinurad 400 mg Fed (Site 1 and Site 2, Lot A) (Experimental): Day 1: Lesinurad 400 mg (Site 1 or Site 2, Lot A) Day 5: Lesinurad 400 mg (Site 1 or Site 2, Lot A)
  Interventions: Drug: Lesinurad 400 mg (Site 1); Drug: Lesinurad 400 mg (Site 2, Lot A)
- Lesinurad 400 mg Fasted (Site 1 and Site 2, Lot B) (Experimental): Day 1: Lesinurad 400 mg (Site 1 or Site 2, Lot B) Day 5: Lesinurad 400 mg (Site 1 or Site 2, Lot B)
  Interventions: Drug: Lesinurad 400 mg (Site 1); Drug: Lesinurad 400 mg (Site 2, Lot B)
- Lesinurad 400 mg Fed (Site 1 and Site 2, Lot B) (Experimental): Day 1: Lesinurad 400 mg (Site 1 or Site 2, Lot B) Day 5: Lesinurad 400 mg (Site 1 or Site 2, Lot B)
  Interventions: Drug: Lesinurad 400 mg (Site 1); Drug: Lesinurad 400 mg (Site 2, Lot B)

INTERVENTIONS:
Drug: Lesinurad 400 mg (Site 1)
Drug: Lesinurad 400 mg (Site 2, Lot A)
  Arms: Lesinurad 400 mg Fasted (Site 1 and Site 2, Lot A); Lesinurad 400 mg Fed (Site 1 and Site 2, Lot A)
Drug: Lesinurad 400 mg (Site 2, Lot B)
  Arms: Lesinurad 400 mg Fasted (Site 1 and Site 2, Lot B); Lesinurad 400 mg Fed (Site 1 and Site 2, Lot B)

SUMMARY:
This study will assess the relative bioavailability of lesinurad tablets, manufactured at two different sites.

DETAILED DESCRIPTION:
A change in manufacturing site of lesinurad tablets has been implemented. This study is intended to evaluate the clinical comparability of lesinurad tablets manufactured at the two different sites by assessing relevant clinical Pharmacokinetics (PK) parameters.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a body weight ≥ 50 kg (110 lbs) and a body mass index (BMI) ≥ 18 and ≤ 40 kg/m2.
* Subject has a Screening sUA value ≤ 7.0 mg/dL.
* Subject is free of any clinically significant disease that requires a physician's care and/or would interfere with study evaluations or procedures.
* Subject has no clinically relevant abnormalities in vital signs, ECG, physical examination or safety laboratory values per the Investigator's judgment.

Exclusion Criteria:

* Subject has a history or clinical manifestations of significant metabolic, hematological, pulmonary, cardiovascular, gastrointestinal, neurologic, hepatic, renal, urological, or psychiatric disorders.
* Subject has a history or suspicion of kidney stones.
* Subject has a history of asthma.
* Subject has undergone major surgery within 3 months prior to Day 1.
* Subject has donated blood or experienced significant blood loss (> 450 mL) within 12 weeks prior to Day 1 or gave a plasma donation within 4 weeks prior to the Screening visit.
* Subject has inadequate venous access or unsuitable veins for repeated venipuncture.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2013-11; Primary Completion 2014-04 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
PK profile of lesinurad from plasma | Day 1 and Day 5
  PK endpoints in terms of maximum observed concentration (Cmax); time of occurrence of maximum observed concentration (Tmax); area under the plasma concentration time curve (AUC); and apparent terminal half-life (t1/2).

SECONDARY OUTCOMES:
Incidence of Adverse Events | 5 weeks
  Changes in Laboratory, Electrocardiogram and Vital Signs Parameters

CONTACTS AND LOCATIONS:
Overall Officials: J. Hall, MD, Study Director — Ardea Biosciences, Inc.
Locations (1):
- Glendale, California, United States